CLINICAL TRIAL: NCT06056362
Title: Evaluation of Biodistribution, Dosimetry, Diagnostic Ability, and Safety of Al18F-NOTA-LM3 in Patients With Well-differentiated Neuroendocrine Tumors, and Comparison With 68Ga-DOTATATE and 68Ga-NODAGA-LM3: A Prospective, Single-center, Double-blinded Study
Brief Title: Comparison of Al18F-NOTA-LM3 With 68Ga-DOTATATE and 68Ga-NODAGA-LM3 PET/CT in Patients With Well-differentiated Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ALFLM3NET
Record Dates: First submitted 2023-03-19; First posted 2023-09-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-09

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The images of patients will be reviewed by 2 experienced nuclear medicine physicians and they will be masked to all patients' clinical information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Al18F-NOTA-LM3 and 68Ga-DOTATATE group (Experimental): Patients will perform an Al18F-NOTA-LM3 PET/CT as well as a 68Ga-DOTATATE PET/CT.
  Interventions: Diagnostic Test: Al18F-NOTA-LM3; Diagnostic Test: 68Ga-DOTATATE
- Arm B: Al18F-NOTA-LM3 and 68Ga-NODAGA-LM3 group (Experimental): Patients will perform an Al18F-NOTA-LM3 PET/CT as well as a 68Ga-NODAGA-LM3 PET/CT.
  Interventions: Diagnostic Test: Al18F-NOTA-LM3; Diagnostic Test: 68Ga-NODAGA-LM3

INTERVENTIONS:
Diagnostic Test: Al18F-NOTA-LM3 — 40 patients will be enrolled in this arm. The first enrolled 8 patients will undergo serial whole-body PET/CT scans at multiple time points (5, 15, 30, 45, 60, and 120 min) after injection of Al18F-NOTA-LM3. The following patients will undergo a whole-body PET/CT scan 60-120 minutes after injection.
  Arms: Arm A: Al18F-NOTA-LM3 and 68Ga-DOTATATE group
Diagnostic Test: 68Ga-DOTATATE — All patients in arm A will undergo a whole-body PET/CT scan 40-60 minutes after injection of 68Ga-DOTATATE. 68Ga-DOTATATE PET/CT and Al18F-NOTA-LM3 PET/CT should be performed within a week and the interval between the two scans at least 24h.
  Arms: Arm A: Al18F-NOTA-LM3 and 68Ga-DOTATATE group
Diagnostic Test: Al18F-NOTA-LM3 — 40 patients will be enrolled in this arm. All patients will undergo a whole-body PET/CT scan 60-120 minutes after injection.
  Arms: Arm B: Al18F-NOTA-LM3 and 68Ga-NODAGA-LM3 group
Diagnostic Test: 68Ga-NODAGA-LM3 — All patients in arm B will undergo a whole-body PET/CT scan 40-60 minutes after injection of 68Ga-NODAGA-LM3. 68Ga-NODAGA-LM3 PET/CT and Al18F-NOTA-LM3 PET/CT should be performed within a week and the interval between the two scans at least 24h.
  Arms: Arm B: Al18F-NOTA-LM3 and 68Ga-NODAGA-LM3 group

SUMMARY:
This prospective, single-center, double-blinded study investigates the biodistribution, dosimetry, safety, and diagnostic ability of Al18F-NOTA-LM3 in patients with well-differentiated neuroendocrine tumors. And compares the diagnostic ability of Al18F-NOTA-LM3 with 68Ga-DOTATATE PET/CT and 68Ga-NODAGA-LM3 PET/CT. Clinical management will also be compared using different imaging modalities.

DETAILED DESCRIPTION:
Somatostatin receptors (SSTR), especially SSTR subtype 2 (SSTR2), are highly expressed in well-differentiated neuroendocrine tumors (NETs). Radiolabeled somatostatin analogs, including 68Ga-DOTATATE, are widely used for NET imaging and play essential roles in primary tumor seeking, staging, as well as management. SSTR antagonists have recently emerged as another type of somatostatin analog and showed better performance than analogs. Our previous studies exhibited better diagnostic efficacy of 68Ga-DOTA-LM3, 68Ga-DOTA-JR11, and 68Ga-NODAGA-LM3 compared to 68Ga-DOTATATE, especially liver metastasis.

18F-labeled radiotracers have shown several advantages compared to 68Ga-labelled tracers, including increased cyclotron production, lower positron energy, and longer half-life when compared to 68Ga, theoretically to the benefit of image quality. The purpose of this study is to investigate the biodistribution, safety, and diagnostic ability of Al18F-NOTA-LM3 in patients with well-differentiated neuroendocrine tumors. And compare the diagnostic ability of Al18F-NOTA-LM3 with 68Ga-DOTATATE PET/CT and 68Ga-NODAGA-LM3 PET/CT. Clinical management related to imaging will also be compared.

Patients with histologically confirmed well-differentiated neuroendocrine tumors (G1 and G2) will be recruited in this study. All patients will be randomized into two arms (A and B): Patients in arm A performed Al18F-NOTA-LM3 and 68Ga-DOTATATE. Patients in arm B performed Al18F-NOTA-LM3 and 68Ga-NODAGA-LM3. The first eight patients will undergo serial PET scans at 5, 15, 30, 45, 60, and 120 min after injection of Al18F-NOTA-LM3. The following patients will perform a whole-body PET/CT scan at 60-90 minutes after injection of Al18F-NOTA-LM3. All patients a whole-body PET/CT scan at 40-60 minutes after administering 68Ga-DOTATATE or 68Ga-NODAGA-LM3. For each patient, the two pet scans should be done within a week and the interval between the two scans should be at least 24h in case of mutual interference.

The images were reviewed by 2 experienced nuclear medicine physicians who were masked to all patients' clinical information. The results were based on consensus, with any discrepant result resolved by a consensus image interpretation by a third senior physician.

The biodistribution, dosimetry, safety, and diagnostic ability of Al18F-NOTA-LM3 will be explored. The diagnostic ability of Al18F-NOTA-LM3 with 68Ga-DOTATATE PET/CT and 68Ga-NODAGA-LM3 PET/CT will be compared. We will also compare the clinical management using different imaging modalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years.
* Histologically proven, well-differentiated, NETs (G1 or G2).
* No long-acting somatostatin analog treatment within 4 weeks.
* No PRRT treatment within 8 weeks.

Exclusion Criteria:

* Combined with other types of tumors.
* Severe liver or renal dysfunction (ALT/AST≥5 ULN, GFR<30ml/min).
* Active infection.
* Pregnant or breast-feeding women.
* Inability to perform PET/CT scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-03-27 (Estimated); Study Completion 2025-03-27 (Estimated)

PRIMARY OUTCOMES:
Safety of Al18F-NOTA-LM3 | From radiotracer injection to 24 hours post-injection.
  Adverse effects were recorded according to CTCAE (version 5.0) after radiotracer injection and PET scan.
Detection rate of Al18F-NOTA-LM3 on per-patient basis | From study completion to 6 months after completion.
  Percentage of patients with lesions detected on Al18F-NOTA-LM3 PET/CT.
SUVmax of lesions detected on Al18F-NOTA-LM3 PET/CT | From study completion to 6 months after completion.
  The tracer uptake is quantified using maximal standard uptake value (SUVmax) by drawing a 3-dimensional region of interest.
Detection rate of 68Ga-DOTATATE on per-patient basis | From study completion to 6 months after completion.
  Percentage of patients with lesions detected on 68Ga-DOTATATE PET/CT.
SUVmax of lesions detected on 68Ga-DOTATATE PET/CT | From study completion to 6 months after completion.
  The tracer uptake is quantified using maximal standard uptake value (SUVmax) by drawing a 3-dimensional region of interest.
Detection rate of 68Ga-NODAGA-LM3 on per-patient basis | From study completion to 6 months after completion.
  Percentage of patients with lesions detected on 68Ga-NODAGA-LM3 PET/CT.
SUVmax of lesions detected on 68Ga-NODAGA-LM3 PET/CT | From study completion to 6 months after completion.
  The tracer uptake is quantified using maximal standard uptake value (SUVmax) by drawing a 3-dimensional region of interest.

SECONDARY OUTCOMES:
SUVmax of normal organs | From study completion to 6 months after completion.
  The biodistribution of Al18F-NOTA-LM3 will be evaluated in the following organs: pituitary gland, parotids, thyroids, lungs, blood pool, liver, spleen, pancreas (head and uncinate process), gallbladder, stomach, small intestine, kidneys, and adrenal glands. SUVmax of these organs were measured and recorded.
Absorbed dose of target organs | From study completion to 6 months after completion.
  Absorbed dose of target organs were calculated using HERMES software.

CONTACTS AND LOCATIONS:
Overall Officials: Meixi Liu, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu M, Zhang Y, Yan X, Zhang H, Ren C, Huang Z, Cheng Y, Xu Q, Li Y, Jia R, Zhu W, Huo L. Assessment of the diagnostic efficacy and clinical significance of [18F]AlF-NOTA-LM3 PET/CT in patients with well-differentiated neuroendocrine tumors. Eur J Nucl Med Mol Imaging. 2026 Jan;53(2):954-967. doi: 10.1007/s00259-025-07484-9. Epub 2025 Aug 5. PMID 40762797
- [Derived] Liu M, Ren C, Zhang H, Zhang Y, Huang Z, Jia R, Cheng Y, Bai C, Xu Q, Zhu W, Huo L. Evaluation of the safety, biodistribution, dosimetry of [18F]AlF-NOTA-LM3 and head-to-head comparison with [68Ga]Ga-DOTATATE in patients with well-differentiated neuroendocrine tumors: an interim analysis of a prospective trial. Eur J Nucl Med Mol Imaging. 2024 Oct;51(12):3719-3730. doi: 10.1007/s00259-024-06790-y. Epub 2024 Jun 15. PMID 38878175